CLINICAL TRIAL: NCT00019461
Title: A Phase II Trial of Orally Administered CAI for Patients With Persistent or Refractory Epithelial Ovarian Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Brief Title: Carboxyamidotriazole in Treating Patients With Refractory or Recurrent Ovarian Epithelial, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066216; NCI-98-C-0012; NCI-T97-0112; NCT00001682 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2003-06

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — carboxyamido-triazole; Drug Therapy

INTERVENTIONS:
Drug: carboxyamidotriazole
Drug: chemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of carboxyamidotriazole in treating patients with refractory or recurrent ovarian epithelial, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical outcome in patients with ovarian epithelial, fallopian tube, or primary peritoneal cancer treated with carboxyamidotriazole.

OUTLINE: Patients receive oral carboxyamidotriazole daily beginning on day 1. Treatment continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 19-40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed refractory or recurrent ovarian epithelial, fallopian tube, or primary peritoneal cancer
* Measurable disease by physical exam, radiography, peritoneoscopy, or laparoscopy

  * No more than 4 weeks since prior peritoneoscopy
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 4 months

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL AND/OR
* Hematocrit at least 27%

Hepatic:

* SGOT/SGPT no greater than 3 times upper limit of normal
* Bilirubin normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No history of symptomatic cardiac dysrhythmias requiring medication
* At least 6 months since prior myocardial infarction
* No unstable or newly diagnosed angina

Pulmonary:

* No obstructive lung disease requiring oxygen therapy

Other:

* Not pregnant or nursing
* HIV negative
* Must be able to take oral medication
* No concurrent medical condition (e.g., impending bowel obstruction)
* No grade 2 or greater residual peripheral neuropathy
* No active infection
* No other prior or concurrent invasive malignancy within the past 5 years
* No history of acute visual loss other than that associated with retinal detachment

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior cytokine therapy
* No concurrent cytokine therapy to maintain WBC count

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas, carboplatin, or mitomycin)
* No other concurrent chemotherapy

Endocrine therapy:

* At least 4 weeks since prior hormonal therapy
* No concurrent corticosteroids at doses greater than physiological replacement doses
* No concurrent hormonal therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No more than 3 prior treatment regimens
* At least 1 week since prior systemic antibiotics for infection
* No chronic antifungal treatment with antimycotic imidazoles
* No concurrent alternative therapies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-04; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahrukh Hussain, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Hussain MM, Kotz H, Minasian L, Premkumar A, Sarosy G, Reed E, Zhai S, Steinberg SM, Raggio M, Oliver VK, Figg WD, Kohn EC. Phase II trial of carboxyamidotriazole in patients with relapsed epithelial ovarian cancer. J Clin Oncol. 2003 Dec 1;21(23):4356-63. doi: 10.1200/JCO.2003.04.136. PMID 14645425